CLINICAL TRIAL: NCT01396460
Title: Respiratory Quotient in Post Roux-en-Y Gastric Bypass Patients
Acronym: RQ
Status: Completed | Type: Observational
Sponsor: Gastrocirurgia, Brazil (Other)
Responsible Party: Principal Investigator, Silvia Leite Faria, Silvia Leite Faria , MSc, RD, Gastrocirurgia, Brazil
Other Study IDs: NCT01231087
Record Dates: First submitted 2011-07-15; First posted 2011-07-18 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Morbid Obesity
Keywords: respiratory quotient; fat oxidation; morbid obesity; bariatric; Bariatric Surgery
MeSH Terms: conditions — Obesity, Morbid | interventions — Breakfast

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- bariatric patients: Bariatric post operative patients were compared with morbid obese population
  Interventions: Other: breakfast (a chicken sandwich with juice)
- control group: morbid obese population

INTERVENTIONS:
Other: breakfast (a chicken sandwich with juice) — patients received a breakfast after de initial measurement
  Groups: bariatric patients

SUMMARY:
Through the values of respiratory quotient (RQ) it is possible to estimate the utilization of energy substrates by the body, or if there is a higher or lower fat oxidation. Experimental and clinical studies have shown that after Roux-en-Y Gastric Bypass (RYGBP) there is a decrease in the values of RQ, which may be associated with increased lipid oxidation in the postoperative period.

Diet Induced Thermogenesis (DIT) is an important part of Total Energy Expenditure. We would like to know how it functions among RYGBP patients.

The purpose of this study is to evaluate the RQ and DIT of patients in the post operative phase and compare the result with a control group consisting of morbid obese population.

ELIGIBILITY:
Inclusion Criteria (bariatric patients post-op)

* With more than 1 year after surgery
* Consent given to participate

Exclusion Criteria:

* Pregnant women
* Malnourished patients (anemia)
* Tiroid disorders without treatment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bariatric post operative population
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Diet Induced Thermogenesis | 20min after standard meal
  To examine the possible changes in the thermic effect of food, the patients received a standard meal. They then repeated the test 20 minutes after eating to obtain a reading of the metabolic rate by considering the DIT and RQ in the postprandial period. DIT was calculated as the difference between post prandial metabolic rate and RMR.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrocirurgia de Brasilia, Brasília, Federal District, Brazil